CLINICAL TRIAL: NCT07179822
Title: Can MEP Conditioning Improve Corticospinal Recruitment of Motoneurons in Chronic Cervical SCI?
Brief Title: Motoneuron Recruitment and Motor Evoked Potential Up-Conditioning (MEP) in Spinal Cord Injury (SCI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Northwestern University (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Aiko Thompson, Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00145581; 1R21HD118383 (NIH)
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries and Disorders (SCI/D); Spinal Cord Injury
Keywords: Movement Disorders; Rehabilitation Studies
MeSH Terms: conditions — Spinal Cord Injuries; Disease; Movement Disorders | interventions — Evoked Potentials, Motor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motor Evoked Potential (MEP) Operant Conditioning (Experimental): This intervention requires 6 baseline visits and 24 intervention visits, each of which is approximately 1.5 hours.
  Interventions: Behavioral: Motor Evoked Potential (MEP) Operant Conditioning

INTERVENTIONS:
Behavioral: Motor Evoked Potential (MEP) Operant Conditioning — Operant conditioning is a method to induce behavioral learning based on the consequence (reward) of the behavior. With operant conditioning of the motor evoked potential (MEP), the neuronal excitability and behavior of the corticospinal pathway that involves production of MEP is targeted and trained (i.e., up-trained with up-conditioning). The individual is rewarded only for changing the target muscle's MEP size without changing background muscle activity. Since MEP size reflects the corticospinal excitability at or just before the time of stimulation, during MEP up-conditioning trials, the individual is urged to increase the corticospinal excitability for the target muscle.

SUMMARY:
The purpose of this research study is to examine the effect of a brain stimulation training to improve the function of brain-spinal cord- muscle connections. Because brain-to-muscle pathways are very important in our movement control, restoring function of these pathways may improve movement problems after injuries. Spinal cord injury causes damage to the brain-to-muscle connection. However, when the injury is "incomplete", there is a possibility that some of the brain-to-muscle pathways are still connected and may be trained to improve movement function. For examining brain-to-muscle pathways, investigators use a transcranial magnetic stimulator. Investigators hope that the results of this research study will help us develop new treatments for people who have movement disabilities. This study will require about 42 visits over the first 14 weeks, and another 6 visits over an additional 3 months. Each visit will take about 1 ½ hours.

DETAILED DESCRIPTION:
Regaining arm/hand function is one of the top priorities of individuals with tetraplegia and is a challenging problem, partly due to the complex nature of upper limb motor function. Through mass practice and conventional therapy, functions can be restored partially, likely through compensation rather than induction of relevant corticospinal plasticity. In such cases, corticospinal recruitment of motoneurons and resulting muscle activation could remain impaired and continue to limit function recovery. In people with incomplete SCI, voluntary activation of the muscles below the injury level is often diminished, due at least partly to impaired motor unit behaviors. Abnormal motoneuron recruitment and motor unit firing, also found in other CNS disorders, would certainly hinder effective production of motor functions. Thus, to enhance upper limb motor rehabilitation beyond what conventional therapy has been able to achieve, a method to improve corticospinal recruitment of a targeted pool of motoneurons would be needed. Here, investigators hypothesize that wrist extensor MEP up-conditioning can improve forearm motor functions in people with cervical SCI by increasing the corticospinal excitability and improving corticospinal recruitment of wrist extensor motoneurons.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 yrs old)
* a history of injury to spinal cord at or above C6
* neurologically stable (>1 year post SCI)
* medical clearance to participate
* weak wrist extension at least unilaterally
* expectation that current medication will be maintained without change for at least 3 months.

  * Stable use of anti-spasticity medication (e.g., baclofen, diazepam, tizanidine) is accepted. (Because only neurologically stable subjects will enter this study, medication changes will be unlikely.)
  * In participants with bilateral wrist extension weakness in whom Extensor Carpi Radialis (ECR) MEP can be elicited in both arms, the more severely impaired arm is studied. In participants with unilateral wrist weakness or in participants with bilateral wrist weakness in whom an ECR MEP can be elicited in only one arm, that arm is studied.

Exclusion Criteria:

* motoneuron injury
* unstable medical condition
* cognitive impairment (because the studied intervention is a learning-based intervention)
* a history of epileptic seizures
* a pre-existing or confounding neurological condition (e.g., history of MS, Stroke, Parkinson's disease)
* metal implants in the cranium
* implanted biomedical device in or above the chest (e.g., a cardiac pacemaker, cochlear implant)
* no measurable MEP elicited in the ECR
* inability to produce any voluntary ECR EMG activity
* extensive use of functional electrical stimulation to the arm on a daily basis (as it may interfere with or augment the effects of MEP conditioning itself)
* pregnancy (due to changes in posture and potential medical instability)
* inability or unwillingness of subject or legal guardian/representative to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in the size of the Motor Evoked Potential (MEP) from baseline to final conditioning sessions. | Baseline (average of 6 sessions over 2 weeks) and final phase (average of sessions 19-24 over weeks 7-8 of intervention)
  MEP from each session is expressed as the percent of the initial MEP size (average MEP size from the 6 baseline sessions). The final MEP size is the fitted estimate of the MEP size at the end of 24 intervention sessions. MEP size is a measurement of the integrity of the corticospinal tract.
Change in Spinal Cord Independence Measure--version III (SCIM III) score | Baseline (Week 0), mid-intervention (Week 5, after session 12), post-intervention (Week 9, after session 24), and follow-up at 1 month (Week 13) and 3 months (Week 21) post-intervention.
  To measure basic functional independence, we will use the most recent version of the SCIM (SCIM III), which is self-reported and comprises 19 items in three sub-scales: (1) self-care (6 items, subscore 0-20); (2) respiration and sphincter management (4 items, sub-score 0-40); and (3) mobility (9 items, subscore 0-40). The total score ranges from 0-100. The items are weighted in terms of their presumed clinical relevance. SCIM score will be used for calculation of MCID.

CONTACTS AND LOCATIONS:
Overall Officials: Aiko Thompson, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No